CLINICAL TRIAL: NCT07337889
Title: Conceptualizing Borderline Personality Disorder as a Relationship Use Disorder
Acronym: TLUR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL24_0194
Record Dates: First submitted 2025-12-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-07

CONDITIONS: Borderline Personality Disorder; Borderline Personality Disorder (BPD); Bipolar Disorder (BD)
Keywords: borderline personality disorder; relationship-use disorder
MeSH Terms: conditions — Borderline Personality Disorder; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with borderline personality (Experimental): Patients with borderline personality disorder without bipolar disorder
  Interventions: Other: Relationship-use questionnaire
- Patients with bipolar disorder (Experimental): patients with bipolar disorder without borderline personality disorder
  Interventions: Other: Relationship-use questionnaire
- Healthy controls (Experimental): Healthy controls (i.e. without psychiatric disorders), from the general population
  Interventions: Other: Relationship-use questionnaire

INTERVENTIONS:
Other: Relationship-use questionnaire — Questionnaire adapted from the 'Substance Use Disorders' section of the DSM-5: Disorder related to the use of close relationships

SUMMARY:
This study aims to explore a novel conceptualization of Borderline Personality Disorder (BPD) as a "Relationship Use Disorder." The research proposes that BPD shares key features with behavioral addictions, specifically addiction to interpersonal relationships. The study builds upon previous findings suggesting that individuals with BPD experience intense emotional dysregulation, including negative self-perception, shame, and a compulsive need for external validation. This addiction to relationships, much like substance use disorders, is thought to contribute significantly to the difficulties faced by these individuals, including interpersonal conflicts, self-destructive behaviors, and emotional instability.

The study seeks to demonstrate that the relational difficulties central to BPD meet the diagnostic criteria for addiction as defined by the DSM-5. It will also explore how these relational struggles are mediated by dysfunctional self-perception and whether they are linked to behaviors such as compulsive sexual behaviors (CSBD) or suicidal tendencies. Additionally, the research will investigate the relationship between addiction to relationships and neurobiological factors, including endorphin levels, in individuals with BPD compared to those with bipolar disorder and healthy controls. The hypothesis is that individuals with BPD will exhibit higher levels of relationship addiction, with this addiction being tied to their perception of self-worth and emotional experiences in relationships.

This innovative approach aims to refine the understanding of BPD, reduce stigma, and improve treatment strategies by providing scientific evidence supporting the conceptualization of BPD as a "Relationship Use Disorder."

ELIGIBILITY:
Inclusion Criteria:

* General : aged 18-45
* Specific :
* Borderline personality disorder (BPD)assessed by SCID, without bipolar disorder
* Bipolar disorder (assessed by SCID), without BPD (evaluated by SCID)
* Healthy controls with no psychiatric disorders (screened by SCID).

Exclusion Criteria:

* Psychotic disorders (evaluated by SCID)
* lack of informed consent
* Not affiliated with social security
* Under judicial or administrative confinement or involuntary hospitalization
* Protected by law (e.g., under guardianship)
* Pregnancy or breastfeeding
* Inability to understand, speak, or write in French
* Inability to understand the study's purpose or methodology
* Excluded from another study during the exclusion period
* Participants who have received over €6000 in annual indemnities
* For Bipolar Participants (without BPD) : Current moderate or severe depressive episode (BDI score > 18) or Current hypomanic/manic episode (YMRS < 12)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Relational Addiction | Measured at baseline
  Using the experimental relationship-use questionnaire based on the DSM-5 Substance Use Disorder items among patients with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD, and healthy controls.

SECONDARY OUTCOMES:
Function Acquisition Speed Test (FAST) | Measured at baseline
  Administer the Function Acquisition Speed Test (FAST) to measure how quickly individuals learn associations between stimuli and responses, focusing on emotional biases related to self (e.g., feelings of unworthiness, ridicule) and others (e.g., dependency, validation). The aim is to assess the intensity of emotional biases in BPD patients compared to BD patients and healthy controls.
Visual Analogue Scale (VAS) for Perceived Alignment with BPD | Measured at baseline
  After viewing an educational video explaining Borderline Personality Disorder (BPD) as relational addiction, assess how participants perceive the alignment of their personal experiences with BPD traits, using a Visual Analogue Scale (VAS) ranging from 0 to 10.
Love Addiction Inventory (LAI) | Measured at baseline
  Using the Love Addiction Inventory (LAI), a 24-item self-report scale, to measure symptoms of love addiction. Participants rate their responses on a 5-point Likert scale, with higher scores indicating greater levels of love addiction symptoms, among patients with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD.
Beta-Endorphin Levels | Measured at baseline
  valuate the correlation between beta-endorphin levels and the dimension of relational addiction among patients with BPD, BD, and healthy controls
Dysfunctional Self-Perception and Related Indicators (SES) | Measured at baseline
  Assessing dysfunctional self-perception and its associated indicators-including feelings of emptiness - among BPD group, BD group and HC group, using :
  * Subjective Emptiness Scale (SES): An 8-item self-report scale measuring feelings of inner emptiness. Higher scores indicate greater perceived emptiness.
Dysfunctional Self-Perception and Related Indicators (RSES) | Measured at baseline
  Assessing dysfunctional self-perception and its associated indicators-including self-esteem-among BPD group, BD group and HC group, using :
  - Rosenberg Self-Esteem Scale (RSES): A 10-item self-report scale assessing global self-worth. The total score ranges from 0 to 30, with higher scores indicating higher self-esteem.
Dysfunctional Self-Perception and Related Indicators (ESS) | Measured at baseline
  Assessing dysfunctional self-perception and its associated indicators-including shame,-among BPD group, BD group and HC group, using :
  - Experience of Shame Scale (ESS): A 25-item self-report scale covering eight domains of shame experiences, including personal habits, interpersonal behaviors, and body image. Higher scores reflect greater shame experiences.
Dysfunctional Self-Perception and Related Indicators (VAS) | Measured at baseline
  Assessing dysfunctional self-perception and its associated indicators-including shame,-among BPD group, BD group and HC group, using :
  - Visual Analog Scale (VAS) for Psychological Pain: Participants mark a point on a 10 cm line that represents their current level of psychological pain. Higher values indicating greater psychological pain.
Painful Experiences Related to the Relational Object (MSR) | Measured at baseline
  Assessing the impact of painful relational experiences, focusing on rejection sensitivity, among patients diagnosed with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD, and healthy controls (HC), using :
  - Rejection Sensitivity Scale (MSR): A 9-item self-report scale assessing the level of anxiety and likelihood of perceiving rejection in various interpersonal situations. Higher scores indicate greater sensitivity to rejection.
Painful Experiences Related to the Relational Object (ESUL) | Measured at baseline
  Assessing the impact of painful relational experiences, focusing on loneliness, among patients diagnosed with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD, and healthy controls (HC), using :
  - University of Laval Loneliness Scale (ESUL): A 20-item self-report scale measuring perceived loneliness in adults. The scale assesses both emotional and social loneliness. Higher scores indicate greater loneliness.
Painful Experiences Related to the Relational Object (RSQ) | Measured at baseline
  Assessing the impact of painful relational experiences, focusing on attachment styles, among patients diagnosed with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD, and healthy controls (HC), using :
  - Relationship Scale Questionnaire (RSQ): A 30-item self-report scale evaluating attachment styles and relational anxiety. Higher scores reflect more insecure attachment styles.
Compulsive Sexual Behavior Disorder | Measured at baseline
  Assessing the severity of compulsive sexual behaviors (CSBD) among patients with Borderline Personality Disorder (BPD) without Bipolar Disorder (BD), those with BD without BPD, and healthy controls (HC), using :
  - Compulsive Sexual Behavior Scale (CSBD-19): a 19-item self-report scale that assesses the severity of compulsive sexual behaviors, following the diagnostic guidelines of the ICD-11. The scale evaluates key dimensions of CSBD, including control, salience, relapse, dissatisfaction, and negative consequences. Participants rate the frequency and impact of their sexual behaviors and impulses on a 5-point Likert scale. Higher scores indicate more severe compulsive sexual behavior.
Non-Relational Addictive Propensity | Measured at baseline
  Assessment of Non-Relational Addictive Behaviors in Patients with Borderline Personality Disorder (BPD), Bipolar Disorder (BD), and Healthy Controls (HC), using substance use disorder criteria.
  Participants will be screened for a range of substances (e.g., alcohol, opioids, stimulants) and will be asked about the frequency, quantity, and impact of substance use in their life.
Suicidal Tendencies | Measured at baseline
  Assessment of Suicidal Tendencies in Patients with Borderline Personality Disorder (BPD), Bipolar Disorder (BD), and Healthy Controls (HC), using :
  * Columbia-Suicide Severity Rating Scale (C-SSRS): The C-SSRS is a clinician-administered assessment tool designed to measure the severity and frequency of suicidal and para-suicidal behaviors. The scale includes questions about lifetime suicidal ideation, recent suicidal ideation, and behaviors, including planning, attempts, and self-injurious actions.